CLINICAL TRIAL: NCT01034475
Title: An Open Label, Dose-Escalation Study to Evaluate Safety, Tolerability, Maximum Tolerated Dose (MTD), Efficacy, and Pharmacokinetics (PKs) of CPI-613 Given Twice Weekly for Three Consecutive Weeks in Patients With Advanced Hematologic Malignancies
Brief Title: Study to Evaluate Safety, Tolerability, Maximum Tolerated Dose (MTD), Efficacy, and Pharmacokinetics (PKs) of CPI-613 Given Twice Weekly for Three Consecutive Weeks in Patients With Advanced Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00012124; CCCWFU 29109 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Advanced Hematologic Malignancies
Keywords: acute myeloid leukemia; acute lymphoblastic leukemia; multiple myeloma; chronic myeloid\ leukemia in blast phase
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Multiple Myeloma | interventions — devimistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CPI-613 (Experimental): CPI-240 mg/m2
  Interventions: Drug: CPI-613

INTERVENTIONS:
Drug: CPI-613 — This is a Phase I open label trial using a 2-stage dose-escalation scheme (single-patient & traditional stages):
  Single-Patient Dose-Escalation Stage: In the single-patient stage, a single patient will be accrued per dose level. The starting dose will be 420 mg/m². Dose level will be escalated (by doubling the previous dose) if there is no toxicity or if the toxicity is grade 1 or less. If toxicity is >Grade 1, the traditional dose-escalation stage will be triggered.
  Traditional Dose-Escalation: All dose escalations conducted in this Traditional Dose-Escalation stage will be escalated according to the modified Fibonacci Dose-Escalation scheme.

SUMMARY:
Chemotherapy resistance is a major cause of death in patients with advanced hematologic malignancies. The proposed novel mechanism of action, non-cross resistance with chemotherapeutic agents currently used in the clinic, and lack of CPI-613-related myelosuppression preclinically and clinically to date make CPI-613 a suitable candidate for phase I clinical trial in these patients. The current trial is one of several clinical trials of CPI-613. Other clinical trials that are conducted in patients with solid tumors have already been initiated.

The primary objective of this study is to determine the safety and MTD of CPI-613 when administered 2x weekly for 3 consecutive weeks.

The secondary objective is to determine the PKs of CPI-613 following IV administration and to observe the anti-tumor effects of CPI-613, if any occur.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically documented relapsed and/or refractory hematologic malignancy
* Karnofsky Performance Status (KPS) of >70%.
* Must be ≥18 years of age.
* Expected survival >1 month.
* Women of child-bearing potential must use accepted contraceptive methods
* No radiotherapy, treatment with cytotoxic agents (except CPI-613), treatment with biologic agents or any anti-cancer therapy within the 3 weeks prior to treatment with CPI-613.

Exclusion Criteria:

* Serious medical illness, such as significant cardiac disease (e.g. symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmia, or New York Heart Association Class III or IV), or severe debilitating pulmonary disease, that would potentially increase patients' risk for toxicity.
* Patients with active central nervous system (CNS) or epidural tumor.
* Any active uncontrolled bleeding, and any patients with a bleeding diathesis (e.g., active peptic ulcer disease).
* Pregnant women, or women of child-bearing potential not using reliable means of contraception.
* Lactating females because the potential of excretion of CPI-613 into breast milk.
* Life expectancy less than 1 month.
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-03; Primary Completion 2013-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
To determine the safety and MTD of CPI-613 when administered 2x weekly for 3 consecutive weeks. | 3 weeks

SECONDARY OUTCOMES:
To determine PKs of CPI-613 following IV administration. | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

REFERENCES:
- [Result] Pardee TS, Lee K, Luddy J, Maturo C, Rodriguez R, Isom S, Miller LD, Stadelman KM, Levitan D, Hurd D, Ellis LR, Harrelson R, Manuel M, Dralle S, Lyerly S, Powell BL. A phase I study of the first-in-class antimitochondrial metabolism agent, CPI-613, in patients with advanced hematologic malignancies. Clin Cancer Res. 2014 Oct 15;20(20):5255-64. doi: 10.1158/1078-0432.CCR-14-1019. Epub 2014 Aug 27. PMID 25165100